CLINICAL TRIAL: NCT04212455
Title: Establishing Biobank in a Cohort Study for Hypertensive Patients in Guangdong Province(GDP Study)
Brief Title: A Cohort Study on Biomarkers of Hypertension in Guangdong Province(GDP Study)
Status: Recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019343H(R2)
Record Dates: First submitted 2019-12-24; First posted 2019-12-27 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Hypertension; Cardiovascular Diseases
Keywords: Hypertension; Cardiovascular Diseases; Mortality; Biomarker
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — This study will collect 20 mL whole blood samples from subjects at one or more study visits. The whole blood will be processed to plasma and stored for testing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-interventional study — This is an observational, non-interventional study

SUMMARY:
Hypertension is the most common chronic diseases and a most important risk factor for cardiovascular and cerebrovascular diseases, and also a substantial public health problem. The purpose of the study is to investigate the association between biomarkers and adverse outcomes in patients with hypertension.

DETAILED DESCRIPTION:
Study population includes subjects who are hypertension, of any race or ethnicity, 18 or older years of age, and have provided written informed consent to provide whole blood specimens at one or more study visits.

Physical examination, questionnaire survey and biological sample collection will be conducted at baseline and the incidence of all-cause and cardiovascular mortality will be investigated during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* In accordance with the diagnosis of hypertension (including Blood pressure ≥140/90mmHg and/or taking antihypertensive drugs and/or self-reported hypertension)

Exclusion Criteria:

* <18 years old
* Unsigned informed consent
* Pregnant Women and Lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypertension
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
All-Cause Mortality | From date of inclusion until the date of death from any cause, assessed up to 1 year
  All-cause mortality was confirmed through a combination of hospital medical records, telephone contacts with patients or family members, and death registration at the Guangdong Provincial Center for Disease Control and Prevention.

SECONDARY OUTCOMES:
Cardiovascular Mortality | From date of inclusion until the date of death from any cause, assessed up to 1 year
  Cardiovascular mortality was defined as death attributable to an ischemic cardiovascular cause (including fatal MI, stroke).

OTHER OUTCOMES:
Secondary outcomes of cardiovascular diseases | Through study completion, an average of 1 years
  The number of and the incidence rate of cardiovascular diseases.
Secondary outcomes of cerebrovascular diseases | Through study completion, an average of 1 years
  The incidence rate of cerebrovascular diseases.
Secondary outcomes of kidney | Through study completion, an average of 1 years
  The incidence rate of hypertensive renal injure and end-stage renal disease
others | From date of inclusion until the date of first event, assessed up to 1 year
  Number of participants with reported hospitalization due to other diseases(eg. diabetes， tumor)

CONTACTS AND LOCATIONS:
Overall Officials: Feng Ying-qing, PhD, Study Director — Guangdong Provincial People's Hospital
Locations (2):
- China (2):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Guangdong Cardiovascular Institute, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No